CLINICAL TRIAL: NCT02390778
Title: Reducing Secondary Distress in Violence Researchers: a Randomised Trial of the Effectiveness of Group Debriefings.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Heidi Grundlingh, Research Fellow, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSHTM#8118
Record Dates: First submitted 2015-03-11; First posted 2015-03-18 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Emotional Distress
Keywords: secondary traumatic stress; vicarious trauma; secondary distress
MeSH Terms: conditions — Compassion Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Debrief Group (Experimental): The debrief group participated in 3 consecutive face-to-face group debriefing sessions lasting 1.5-2 hrs each. Each session started with a fun ice-breaker to create a relaxed atmosphere and group cohesion. Session 1 focused on encouraging group participation, discussing primary trauma encountered and emotional reactions to these stories. Session 2 connected current experiences with the group members' own trauma histories and life experiences. The last session focussed on societal and community responses to violence, and employing personal agency to find constructive ways to address violence in communities.
  Interventions: Behavioral: Group Debriefing
- Control Group (Placebo Comparator): The control group was assigned to a leisure activity (film showing), for every session of debriefing undergone by the intervention group. The films were chosen for their light-hearted uplifting content and presented as a fun and relaxing activity.
  Interventions: Behavioral: leisure activity (film showing)

INTERVENTIONS:
Behavioral: Group Debriefing — Group Debriefing involves story-telling, identifying emotional responses to these stories, psycho-education and practical information to normalize group member reactions to a distressing event.
  Arms: Debrief Group
Behavioral: leisure activity (film showing)
  Arms: Control Group

SUMMARY:
The objectives of the study were: To (1) describe the epidemiology of emotional distress experienced by Ugandan violence researchers; to (2) assess the effectiveness of group debriefings in mitigating secondary distress; to (3) assess risk and protective factors. Eligible participants were 59 Ugandan researchers employed by the Good Schools Study (GSS, NCT01678846) to interview children and adults who experienced violence. Recruited participants were randomly assigned to group debriefings (intervention) or film viewing (control). The primary outcome was change in levels of emotional distress.

DETAILED DESCRIPTION:
Background: Secondary distress including emotional distress, vicarious trauma (VT) and secondary traumatic stress (STS) due to exposure to primary trauma victims have been described in helping professionals and in violence researchers. To our knowledge, there are few prevalence studies, and no tailored interventions have been tested to reduce secondary distress in violence researchers.

Objective: To (1) describe the epidemiology of emotional distress experienced by Ugandan violence researchers; to (2) assess the effectiveness of group debriefings in mitigating secondary distress; to (3) assess risk and protective factors.

Methods: An unblinded, individually randomised trial with parallel assignment was conducted. Eligible participants were 59 Ugandan researchers employed by the Good Schools Study (GSS, NCT01678846) to interview children and adults who experienced violence in the district of Luwero, Uganda. 53 researchers agreed to participate and were randomly allocated. The intervention group (n=26) participated in three group debriefings and the control group (n=27) participated in three leisure sessions (film viewing).The primary outcome was change in levels of emotional distress (SRQ-20); secondary outcomes were levels of VT and STS at end-line.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were all 59 Ugandan researchers who had been employed by the GSS.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline Self-Report Questionnaire-20 (SRQ-20) score at 5 weeks | 5 weeks
  The SRQ-20 is a 20 item measure which require simple 'yes' or 'no' responses and was designed as a screening tool for psychological symptoms/emotional distress. It has been widely used and validated in low and middle-income countries as a measure of mental health and wellbeing. The SRQ-20 was modelled as a continuous variable but also a binary variable were the top 33% of the overall distribution was deemed as having a 'high' score indicative of probable emotional distress, consistent with previous research.

SECONDARY OUTCOMES:
Vicarious Trauma Scale (VTS) at 5 weeks | 5 weeks
  The Vicarious Trauma Scale (VTS), an 8 item measure with a 7 point Likert-type scale, has recently been developed and shown to have good psychometric properties for use as a screening tool for vicarious trauma in low resource settings. It is the only publically available screening measure of VT.
Impact of Events Scale-Revised (IES-R) at 5 weeks | 5 weeks
  The Impact of Events Scale-Revised (IES-R)consists of 22 items with a 4 point Likert-type scale widely validated and used to screen for post-traumatic stress disorder (PTSD). It has been used by several studies to measure STS as the theoretical symptomology is similar.
Professional Quality of Life Scale (ProQOL) at 5 weeks | 5 weeks
  The Professional Quality of Life Scale (ProQOL) was developed to screen mental health and other professionals who may experience positive or negative impacts as they help others. Versions of the screening tool have good construct validity with over 200 published papers and it is widely used in research as a measure for STS and related constructs.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Grundlingh, MPH, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Grundlingh H, Knight L, Naker D, Devries K. Secondary distress in violence researchers: a randomised trial of the effectiveness of group debriefings. BMC Psychiatry. 2017 Jun 2;17(1):204. doi: 10.1186/s12888-017-1327-x. PMID 28578682